CLINICAL TRIAL: NCT03225729
Title: Prospective Clinical Trial to Assess the Performance of a Cyto-selective Cryotherapye "CRYOBEAUTY MAINS ET DECOLLETE" Compared With Liquid Nitrogen Cryotherapy in the Treatment of Solar Lentigines in 30 Patients
Brief Title: Assessment of CRYOBEAUTY MAINS ET DECOLLETE Versus Liquid Nitrogen Cryotherapy, in the Treatment of Solar Lentigines
Acronym: CBT-EC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cryobeauty (Industry)
Collaborators: CEISO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-A02179-44
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Solar Lentigo

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CRYOBEAUTY MAINS ET DECOLLETE (Experimental): CRYOBEAUTY MAINS ET DECOLLETE is a new technology conceived to treat solar lentigo.
  One side left, or right of neckline and/or hands is attributed to this device according to randomization protocol.
  Interventions: Device: CRYOBEAUTY MAINS ET DECOLLETE
- Liquid nitrogen (Active Comparator): Liquid nitrogen is a classic cryotherapy device. One side, either left or right of neckline and/or hands are attributed to this device according to randomization protocol.
  Interventions: Device: Liquid nitrogen

INTERVENTIONS:
Device: CRYOBEAUTY MAINS ET DECOLLETE — The intervention lasts up to 6.5 s. The device will be applied on spots <6 mm which are previously selected by the investigator team.
  Arms: CRYOBEAUTY MAINS ET DECOLLETE
Device: Liquid nitrogen — The intervention lasts up to 3 s. The liquid is stored in well-isolated recipients. Each patient has his recipient to avoid contamination. The investigator applies on spots <6 mm a small amount of nitrogen liquid.
  Other Names: Azote médical liquide
  Arms: Liquid nitrogen

SUMMARY:
This study evaluates the performance of new technology "CRYOTHERAPY MAINS ET DECOLLETE" against a classic cryotherapy "Nitrogen Liquid " to treat solar lentigines.

The hands and the neckline will be randomised, either left or right side and treated by two cryotherapy devices:

1. CRYOTHERAPY MAINS ET DECOLLETE is the device under evaluation.
2. Liquid nitrogen is a comparator device.

ELIGIBILITY:
Inclusion Criteria:

* Phototype II to IV
* Presenting solar lentigos on both hands and neck, diameter ≤ 6mm
* Accepting not to expose the body to sunlight or artificial UV rays during the study
* Affiliate to a health insurance plan
* Having undergone a general clinical examination attesting to his / her ability to participate in the study
* Having given written consent

Exclusion Criteria:

* Having carried out aesthetic care (exfoliants, scrubs or self-tanning, manicure, hand care, UV ...) in the month before the start of the study, at the level of the hands and/or neckline.
* Having applied a depigmenting product in the month preceding the start of the study, at the level of the hands and/or neckline.
* Having carried out aesthetic care at a dermatologist (laser, IPL, peeling, depigmenting creams, cryotherapy ...), at the level of the hands and/or neckline, during the last six months
* Dermatosis, autoimmune disease (vitiligo), systemic, chronic or acute disease, or any other disease that may interfere with the treatment or influence the results of the study (people with diabetes, circulatory problems, cold allergies, With Raynaud's syndrome ...)
* Receiving general or local treatment (corticosteroids ...) likely to interfere with the evaluation of the studied parameters.
* Participating in another study or being in an exclusion period from a previous study
* Being incapable of following the requirements of the protocol
* Person protected by law
* Unable to read and write French
* Pregnant woman or woman wishing to be pregnant during the study, or during breastfeeding period
* Women of childbearing age who do not have contraception

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Performance assessment of new cryotherapy device "CRYOTHERAPY MAIN ET DECOLLETE" to treat solar lentigo spots on the hands. | 8 weeks
  Evaluation of CRYOBEAUTY MAINS's performance
  Hexsel scoring:
  1. > Very significant clearance (about 90%); only minor evidence of hyper pigmentation remains
  2. > Significant improvement (about 75%); some signs of hyper pigmentation remains
  3. > Intermediate between marked and slight improvement; about 50% improvement in the appearance of hyper pigmentation
  4. > Some improvement (about 25%); however, significant evidence of hyper pigmentation remains
  5. > Hyperpigmentation has not changed since baseline
  6. > Worse (hyperpigmentation is worse than at baseline)

SECONDARY OUTCOMES:
Performance assessment of CRYOBEAUTY HANDS AND DECOLLETE on the spots of the neckline. | 8 weeks
  Evaluation of CRYOBEAUTY MAINS's performance
  Hexsel scoring:
  1. > Very significant clearance (about 90%); only minor evidence of hyper pigmentation remains
  2. > Significant improvement (about 75%); some signs of hyper pigmentation remains
  3. > Intermediate between marked and slight improvement; about 50% improvement in the appearance of hyper pigmentation
  4. > Some improvement (about 25%); however, significant evidence of hyper pigmentation remains
  5. > Hyperpigmentation has not changed since baseline
  6. > Worse (hyperpigmentation is worse than at baseline)
Evolution of spot's colour | 0 weeks
  Colours assessment: by using Mexameter® MX 18
Evolution of spot's colour | 4 weeks
  Colours assessment: by using Mexameter® MX 18
Evolution of spot's colour | 8 weeks
  Colours assessment: by using Mexameter® MX 18
Pain assessment | 0 weeks
  VAS
Incidence of Treatment-Emergent Adverse Events | 4 weeks
  Adverse events [Safety and Tolerability]
Incidence of Treatment-Emergent Adverse Events | 8 weeks
  Adverse events [Safety and Tolerability]
Assessment of ergonomic and device's readiness | 0 weeks
  Ergonomic and device's readiness questionnaire: 6 QCM questions are given to the participants
Assessment of volunteers feeling (QoL) | 0 weeks
  MelasQoL (Melasma. Quality of Life Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Queille-Roussel, MD, Principal Investigator — Centre de Pharmacologie Clinique Applique a la Dermatologie
Locations (1):
- CPCAD, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided